CLINICAL TRIAL: NCT04306796
Title: 3D Printed Made to Measure Splints for Hand Patients - Pilot Feasibility Study and Socioeconomic Evaluation
Brief Title: 3D Printed Made to Measure Splints for Hand Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-00351;ch20Kaempfen
Record Dates: First submitted 2020-03-04; First posted 2020-03-13 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Splints
Keywords: hand trauma; splint; made to measure; 3D print

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Patients receiving 3D-printed made to measure splints for postoperative or post-traumatic treatment in hand surgical patients
  Interventions: Device: 3D printed splints
- control group (Active Comparator): Patients receiving thermoplastic splints individually adjusted by occupational therapists
  Interventions: Device: Thermoplastic splints

INTERVENTIONS:
Device: 3D printed splints — 3D printed made to measure splints
  Arms: intervention group
Device: Thermoplastic splints — thermoplastic splints individually adjusted by occupational therapists
  Arms: control group

SUMMARY:
This study aims to evaluate the feasibility and possible benefits of 3D-printed made to measure splints for postoperative or post-traumatic treatment in hand surgical patients (intervention group) in comparison to thermoplastic splints individually adjusted by occupational therapists (control group).

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the hand surgical department of the University Hospital Basel
* Patients with hand trauma w/wo the need for hand surgery or patient with planned elective hand surgical intervention
* Indication for immobilization of at least 4 weeks
* Older than 18 years
* Capable of consent
* Informed Consent as documented by signature

Exclusion Criteria:

* Open wounds with tissue loss
* Injury with the need for external fixation
* Younger than 18 years
* Not capable of consent
* Asymmetric deformity or loss of the contra-lateral hand
* Documented hypersensitivity or allergy to Polylactic acid
* Known or suspected non-compliance to agreed treatment measures and/or unexcused nonappearance to hospital appointments
* Drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Change in patient comfort and satisfaction | at 2-5 days after trauma and/or surgery
  questionnaire 1. that will be filled out by the Patient (scale 1-10 and answer text with qualitative assessment)
Change in patient comfort and satisfaction | at 2 weeks of immobilization during a routine control visit
  questionnaire 2. that will be filled out by the Patient (scale 1-10 and answer text with qualitative assessment)
Change in patient comfort and satisfaction | at 6 weeks of immobilization during what is usually the concluding visit of treatment
  questionnaire 3. that will be filled out by the Patient (scale 1-10 and answer text with qualitative assessment)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Plastische, Rekonstruktive, Aesthetische und Handchirurgie,, Basel, Switzerland